CLINICAL TRIAL: NCT02416973
Title: Study of PEMF (Pulsed Electromagnetic Field) Therapy in the Treatment of Persistent Post-Operative Pain Following Lumbar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBI.2015.001
Record Dates: First submitted 2015-03-30; First posted 2015-04-15 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Lumbar Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Sham of Provant (Other): Sham of Provant
  Interventions: Device: Provant
- Active Treatment (Other): Active Provant Treatment
  Interventions: Device: Provant
- Active Treatment with alternative settings (Other): Active Provant Treatment with alternative settings
  Interventions: Device: Provant

INTERVENTIONS:
Device: Provant

SUMMARY:
To demonstrate the analgesic effectiveness of 2 modalities of PEMF treatment compared to sham treatment in patients with persistent pain following lumbar surgery when treatment is administered twice daily over a 60 day period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater than or equal to 22 years.
2. Subject has undergone one or two anatomically successful lumbar back surgeries for the treatment of low back pain.
3. Subject has persistent pain in the low back and/or radiating pain to leg(s) for > 3 months and < 36 months following the most recent surgery. If radiating leg pain is occurring in both legs, one leg, which has the worst Average Pain Intensity over the week prior to the Screening Visit, will be selected as the index leg.
4. Subject has been receiving medication for persistent post-operative low back and/or radiating leg pain, including opioid or non-opioid analgesic medication, and is on a stable analgesic dosing regimen (i.e. the same medications and dosages) for > 30 days prior to the Screening Visit.
5. Average Pain Intensity (calculated as the mean of the daily Average Pain Intensity scores for either back and/or leg) is ≥ 3 and < 9 as measured on Numeric Pain Rating Scale (NPRS) during the 10-day run-in period.
6. Subject has completed a minimum of 80% (8 of 10 possible) of the electronic Patient Reported Outcome (ePRO) assessments during the 10 day run-in period.
7. Subject is able to access an internet browser in the home environment.
8. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol.
9. Female subjects must be post-menopausal, surgically sterile, abstinent, or practicing (or agree to practice) an effective method of birth control if they are sexually active for the duration of the study. (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Exclusion Criteria:

1. Subject has a history of more than two lumbar spine surgeries.
2. Subject requires additional lumbar surgery or surgery of any type prior to Day 75.
3. Subject had disc fusion at any level in the most recent surgery.
4. Subject has received any investigational drug or device within 30 days or 5 half-lives of the drug, whichever is longer, prior to the Screening Visit or is enrolled in another clinical trial.
5. Subject has undergone any local injection into the lumbar spine within 30 days prior to the Screening Visit or within 6 weeks prior to the Screening Visit for long acting lidocaine injection products.
6. Subject has used systemic corticosteroids within 2 months of the Screening Visit.
7. Subject has a history of any uncontrolled medical illness that in the investigator's judgment places the subject at unacceptable risk for receipt of PEMF therapy.
8. Subject has a history of malignancy within the past five years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area and/or localized in situ carcinoma of the cervix.
9. Subject has an ongoing painful condition that in the opinion of the investigator might have a confounding influence on the safety or effectiveness analyses for this study.
10. Subject has a serious psychosocial co-morbidity.
11. Subject has a history of drug or alcohol abuse within one year prior to screening.
12. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
13. Subject consumes an average of > 100 mg oral Morphine Sulfate equivalents per day during the 10 day run-in period.
14. Standard deviation around the mean of the average pain intensity scores during the 10 day run-in period is > 2.0.
15. Subject has a Body Mass Index (BMI) > 38 kg/m2.
16. Subject is currently pregnant or planning on becoming pregnant prior to Day 75.
17. Subject has been previously treated with the PROVANT Therapy System.
18. Subject is in current litigation regarding back pain or is receiving Worker's Compensation.
19. Subject is unwilling or unable to follow study instructions, comply with the treatment regimen, study visits, and ePRO assessments.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - AOC-Research, Birmingham, Alabama
  - Hope Research, Phoenix, Arizona
  - Injury Care Research, Boise, Idaho
  - Rockford Orthopedic, Rockford, Illinois
  - Hope Research_Las Vegas, Las Vegas, Nevada
  - Tarheel Clinical Research, Raliegh, North Carolina
  - Upstate Clinical, Spartanburg, South Carolina
  - Danville Orthopedic, Danville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham of Provant: Sham of Provant
  Provant
- Active Treatment: Active Provant Treatment
  Provant
- Active Treatment With Alternative Settings: Active Provant Treatment with alternative settings
  Provant
Period: Overall Study
Arm/Group | Sham of Provant | Active Treatment | Active Treatment With Alternative Settings
Started | 14 | 13 | 14
Completed | 13 | 10 | 13
Not Completed | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham of Provant | Active Treatment | Active Treatment With Alternative Settings | Total
Number analyzed (Participants) | 14 | 13 | 14 | 41
Age, Continuous [Mean (Full Range); unit: years] | 50.6 [28 to 70] | 54.9 [30 to 81] | 50.2 [30 to 74] | 51.83 [28 to 81]
Gender [Count of Participants; unit: Participants]
  Female | 9 | 5 | 7 | 21
  Male | 5 | 8 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 14 | 41
PainDETECT Questionnaire [Mean (Full Range); unit: units on a scale] — PainDETECT Questionniare (PD-q): a self-reported assessment designed to identify the presence of a neuropathic pain component in subjects with back pain. This was completed by the subject and scored by the research personnel at the Enrollment Visit. Subjects assessment current pain, strongest pain, average pain, areas of pain, course of pain and symptoms (such as burning, tingling, numbness and sensitivity). The scale ranged from 0 to 38 defined as follows: score 0-12 = neuropathic pain component unlikely; 13-18 = result is ambiguous; 19-38 = neuropathic pain component is likely.
  units on a scale | 16.6 [4 to 28] | 14.5 [7 to 19] | 16.1 [2 to 27] | 15.8 [2 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Pain Scores
Description: Numerical Pain Rating Scale (NPRS) was used to score pain at Baseline and at End of Treatment. The Percent change (difference) from Baseline to End of Treatment was calculated. The NPRS is an 11-point scale ranging from scores of 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 60 days
Population: Per protocol population results displayed. This results in a discrepancy in the number of participants provided above. Baseline characteristics include the entire intent to treat population.
Measure: Mean (Standard Deviation); unit: Percent Difference
Arm/Group | Sham of Provant | Active Treatment | Active Treatment With Alternative Settings
Number analyzed (Participants) | 13 | 9 | 13
Percent Difference | -25.6 (24.81) | -40.2 (26.35) | -18.6 (39.47)

ADVERSE EVENTS:
Arm/Group | Sham of Provant | Active Treatment | Active Treatment With Alternative Settings
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 6/13 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham of Provant (N=14) | Active Treatment (N=13) | Active Treatment With Alternative Settings (N=14)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated is not permitted without the prior written consent of sponsor. Such consent may be contingent on sponsor review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.